CLINICAL TRIAL: NCT01736904
Title: A Multicenter, Randomized Phase II Study of Weekly XELIRI Regimen Versus FOLFIRI in the Treatment of Advanced Colorectal Cancer Patients
Brief Title: wXELIRI Versus FOLFIRI Regimen in the Treatment of Advanced Colorectal Cancer Patients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Jin Li, Dr, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: wXELIRI vs FOLFIRI in CRC
Record Dates: First submitted 2012-11-21; First posted 2012-11-29 (Estimated); Last update posted 2012-11-29 (Estimated); Status verified 2012-11

CONDITIONS: Colorectal Cancer
Keywords: advanced colorectal cancer; FOLFIRI; XELIRI
MeSH Terms: conditions — Colorectal Neoplasms | interventions — IFL protocol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- FOLFIRI (Active Comparator): FOLFIRI regimen
  Interventions: Drug: FOLFIRI regimen
- wXELIRI regimen (Experimental): wXELIRI
  Interventions: Drug: wXELIRI regimen

INTERVENTIONS:
Drug: wXELIRI regimen — irinotecan 90mg/m2 D1, capecitabine 1000mg/m2 bid po, D1-5,repeated every 7 days
  Other Names: wXELIRI
  Arms: wXELIRI regimen
Drug: FOLFIRI regimen — irinotecan 180mg/m2 d1,leucovorin 400mg/m2 d1, 5-fluorouracil 400mg/m2 iv, 2.4g/m2 civ 46h, repeated every 2 weeks
  Other Names: FOLFIRI
  Arms: FOLFIRI

SUMMARY:
The aim of this study is to compare weekly-XELIRI(wXELIRI) regimen versus FOLFIRI regimen in the treatment of advanced colorectal cancer patients. The hypothesis is the efficacy of wXELIRI is not less than FOLFIRI with tolerable toxicity.

DETAILED DESCRIPTION:
The combination of irinotecan and fluorouracil drugs regimen is frequently used in patients with advanced colorectal cancer. According to the previous data, higher rate of diarrhea was observed in the combination of irinotecan and capecitabine (XELIRI) regimen, compared to the combination of irinotecan and 5-fluorouracil (FOLFIRI) regimen. However, the modified weekly XELIRI regimen, which was investigated in our previous single armed study, show tolerate toxicities compared with FOLFIRI, without compromising efficacy. It is supposed that wXELIRI regimen is no less less than FOLFIRI regimen in efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Second-line treatment for advanced colorectal cancer,irinotecan was not previously used.
* Age range 18-70 years old
* ECOG performance status 0-1
* Life expectancy of more than 3 months
* Adequate organ function

Exclusion Criteria:

* Previous serious cardiac disease
* History of other malignancies except cured basal cell carcinoma of skin and carcinoma in-situ of uterine cervix
* Pregnant or lactating women
* chronic inflammatory bowel disease or intestinal obstruction
* Serious uncontrolled diseases and intercurrent infection

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2012-05; Primary Completion 2014-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Progression free survival which is calculated from the start of treatment to disease progression or death | eight weeks

SECONDARY OUTCOMES:
Objective response rate which includes complete response(CR) and partial response(PR) participants | eight weeks
  Objective response rate (ORR)= CR(complete response)+PR(partial response)

OTHER OUTCOMES:
Overall survival which is calculated from the start to treatment to the death | eight months

CONTACTS AND LOCATIONS:
Overall Officials: Jin Lin, PhD, MD, Principal Investigator — Fudan University
Locations (1):
- Fudan University Cancer Hospital, Shanghai, Shanghai Municipality, China